CLINICAL TRIAL: NCT07014735
Title: A Single Centre, Placebo-controlled Study to Evaluate the Combined Effect of Hyperglycaemia and a QTc-prolonging Medication on Cardiac Repolarisation in Male and Female Patients With Insulin Resistant Type 2 Diabetes Mellitus (T2DM)
Brief Title: Effect of Hyperglycaemia and Moxifloxacin on QTc Interval in T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richmond Pharmacology Limited (Industry)
Collaborators: Richmond Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: C20032
Record Dates: First submitted 2023-04-18; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Type 2; Hyperglycaemia (Diabetic); QT Interval, Variation in; Torsades de Pointes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Torsades de Pointes | interventions — Glucose; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: The participant will be blinded to the administered medicinal products, but the clinical team will not.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- glucose (controlled hyperglycaemia) and moxifloxacin placebo (Placebo Comparator): Participants will receive glucose (controlled hyperglycaemia) and moxifloxacin placebo on Day 1. On Days 1 and 3 glucose will be administered intravenously and/or orally with the aim of gradually raising glucose concentration to 25-28 mmol/L over the space of an hour. The 25-28 mmol/L glucose level will be maintained for 1 hour. Intravenous glucose rate will be titrated up and down during the first hour as guided by glucose readings on CGMS/VBG. Glucose will be continuously monitored to guarantee concentration levels are maintained stable. At the 2-hour timepoint (H2), intravenous glucose will be terminated, and blood glucose level will be allowed to start reducing.
  Interventions: Drug: glucose
- intravenous glucose in combination with intravenous moxifloxacin (Experimental): intravenous glucose in combination with intravenous moxifloxacin (300 mg infused over 45 minutes) on Day 3
  Interventions: Drug: glucose; Drug: moxifloxacin

INTERVENTIONS:
Drug: glucose — Participants will receive treatments with glucose or matching placebo (please see study design section).
Drug: moxifloxacin — Participants will receive moxifloxacin or matching placebo (please see study design section).
  Arms: intravenous glucose in combination with intravenous moxifloxacin

SUMMARY:
Diabetes is a significant risk factor for sudden cardiac death, with the QTc interval on electrocardiograms (ECGs) often prolonged in diabetic patients due to factors such as hyperglycaemia and insulin resistance. Drugs like moxifloxacin can further exacerbate this effect, especially in those with diabetes. A previous trial on Type 1 diabetes suggested that hyperglycaemia and moxifloxacin have additive effects, prompting an investigation into whether similar effects occur in Type 2 diabetes (T2DM), particularly in individuals with high insulin resistance. This study aims to evaluate whether moxifloxacin-induced QT-prolongation is amplified by elevated blood glucose levels or insulin deficiency in T2DM patients, considering potential differences between sexes. Blood biomarkers will be analysed to understand the underlying molecular mechanisms. The trial will involve at least 24 male and female participants with insulin-resistant T2DM, aged 18 to 64 years, conducted at Richmond Pharmacology Ltd. Participants will receive treatments with glucose, moxifloxacin, and placebos while closely monitored for side effects during an inpatient stay, followed by outpatient appointments.

DETAILED DESCRIPTION:
Diabetes has been established as a key independent risk factor for sudden cardiac death, a common cause of death from cardiovascular disease. The underlying mechanisms for this seem to be complex and multifactorial, but a change in the electrocardiogram (ECG)(which measures the electrical activity of the heart) parameter called QTc interval has been identified as potentially having a significant role. In patients with diabetes, QT interval prolongation is frequently reported. High blood glucose levels (hyperglycaemia) and insulin resistance (the condition where the body does not respond well to insulin) are thought to be important causes. The investigators also know that some drugs e.g., moxifloxacin (a common antibiotic) can prolong the QT interval and this effect can be more pronounced in patients with diabetes.

The investigators have previously conducted a trial on Type 1 diabetes showing that the effects of hyperglycaemia and moxifloxacin were additive. This led to our hypothesis that similar effects might be observed in type 2 diabetes (T2DM), specifically in those with high insulin resistance. Understanding whether the well-established QT-prolongation caused by moxifloxacin is exaggerated by elevated levels of blood glucose alone or by an insulin deficiency is important for evaluating the risk to patients with T2DM and the potential prevention of cardiac complications. The investigators would also like to determine if the effect varies between sexes and gain a comprehensive understanding of the molecular factors driving these differences by analysing blood biomarkers.

This trial will be conducted at Richmond Pharmacology Ltd. involving a minimum of 24 male and female participants with insulin-resistant T2DM, aged 18 to 64 years. The participants will stay in the clinical trials unit, receive treatments with glucose, moxifloxacin, and placebos and will be monitored closely for any side effects. Following the inpatient stay, participants will return to the unit for an outpatient appointment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with stable T2DM. Diagnosis of T2DM confirmed by:

   i. Established diagnosis of T2DM documented on medical records and HbA1c at screening ≥ 48 mmol/mol (6.5%) and ≤ 80 mmol/mol (9.5%). Subjects with HbA1c levels > 80 mmol/mol but ≤ 90 mmol/mol will be considered eligible, subject to approval by an endocrinologist. AND ii. Evidence of high insulin resistance as defined by a HOMA2-IR score within the top quintile of the locally defined cohort, >0.55 (see Appendix 2).
2. 18-64 years (inclusive) of age (at the date of signing informed consent), with a body mass index of 18 to 35 kg/m², inclusive (at screening).
3. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the participant's ability to complete the study as assessed by the Investigator.
4. Stable patients with insulin resistant type 2 diabetes treated with one of the following:

   a. Diet and exercise alone, b. Anti-glycaemic monotherapy on metformin, DPP-4i, pioglitazone, an SU or an SGLT-2i.
5. Able to wash-out anti-glycaemic therapy for ten half-lives prior to dosing or at D-7, whichever is longer, and for the duration of the trial period up to the end of Day 4.
6. Participants must agree to use the following contraceptive requirements for the applicable duration:

   1. Female participants of non-childbearing potential (WNCBP): Defined as either postmenopausal (evidence of menopause based on a combination of amenorrhea for at least one year and increased serum follicle-stimulating hormone (FSH) level [> 30 IU/L]), or surgical sterilization (evidence of hysterectomy and/or bilateral oophorectomy). CONTRACEPTION REQUIRED: None
   2. Female participants of childbearing potential (WOCBP) who anticipate being sexually active with a male during the trial (from one complete menstrual cycle prior to the first drug administration until three months after the last drug administration) *: CONTRACEPTION REQUIRED: Highly effective contraception must start one complete menstrual cycle prior to the first day of dosing and continue until three months after drug administration. Highly effective contraception methods for WOCBP include:

      * Combined i.e. (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation: **

        * Oral
        * Intravaginal
        * Transdermal
      * Progestogen-only hormonal contraception associated with inhibition of ovulation**

        * oral
        * injectable
        * implantable
      * Intrauterine hormone-releasing system (IUS)**
      * Intrauterine device (IUD)
      * Bilateral tubal occlusion
      * Infertile male partner (e.g., vasectomised, permanently sterile following bilateral orchidectomy, or any other documented cause of infertility)
   3. Female participants of childbearing potential (WOCBP) who agree to remain abstinent for the duration of the trial (from one complete menstrual cycle prior to the first drug administration until three months after the last drug administration): CONTRACEPTION REQUIRED: Abstinence (N.B. sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Calendar, symptothermal and post-ovulation methods of contraception are not considered to be equivalent to abstinence).
   4. Male participants, who agree to remain abstinent for the duration of the trial (from first drug administration until three months after the last drug administration): CONTRACEPTION REQUIRED: Abstinence (N.B. sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant). If the situation changes post-dose during the trial, participants must use a condom with or without spermicide.
   5. Male participants, who anticipate being sexually active during the trial period (from first drug administration until three months after the last NIMP administration) with a woman who is either a WOCBP, a woman who is pregnant and/or breast feeding: CONTRACEPTION REQUIRED: From the first day of dosing until the end of the systemic exposure of the trial drug (for this trial this is until the follow-up visit). Acceptable methods are:

      * Male condom with or without spermicide
      * Infertile male (e.g., vasectomised, permanently sterile following bilateral orchidectomy, or any other documented cause of infertility)
7. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any study-related procedures. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. History or clinical evidence of T2DM related secondary complications in particular autonomic neuropathy, cardiac rhythm disturbances, past medical history of syncope and potassium abnormalities.
2. Currently prescribed or used in the last 12 months any form of insulin therapy, or any long half-life diabetic medication that would not wash-out within 7 days.
3. History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study drug (appendicectomy and herniotomy allowed).
4. History or clinical evidence of significant microvascular disease including chronic kidney failure, macular degeneration or any other disease attributed to the microvascular system that in the Investigator's opinion may affect the outcome of the study.
5. Recent hospitalisation due to hypoglycaemia or hyperglycaemia within 28 days before screening.
6. History or clinical evidence of any disease with a specific contraindication to moxifloxacin (hypersensitivity, history of tendon disease related to quinolone treatment, and risk of QT prolongation conditions as below).
7. History of clinically significant syncope.
8. Family history of sudden cardiac death.
9. Clinically significant history or family history of congenital long QT syndrome (e.g., Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada syndrome.
10. History of clinically significant arrhythmias (especially ventricular arrhythmias, atrial fibrillation (AF), recent conversion from AF), or bundle branch block.
11. History of confirmed ischemic heart disease or current angina (including confirmed previous myocardial infarction, previous PCI, or coronary bypass).
12. Conditions predisposing the volunteer to electrolyte imbalances other than T2DM (e.g., altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa, and other endocrine disorders including Cushing's' Addison's', or untreated hypo or hyperthyroidism).
13. ECG abnormalities in the standard 12-lead ECG (at screening, Day -1 or pre-dose of Day 1) and 24-hour 12-lead Holter ECG or an equivalent assessment and/or submaximal exercise test (at screening) which in the opinion of the Investigator will interfere with the ECG analysis.
14. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes. This includes participants with any of the following (at screening,

    Day-1, or pre-dose on Day 1):
    * Sinus node dysfunction.
    * Clinically significant PR (PQ) interval prolongation.
    * Intermittent second or third degree AV block.
    * Incomplete or complete bundle branch block (QRS >110ms).
    * Sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia, any symptomatic arrhythmia except for isolated extra systoles.
    * More than 200 ventricular ectopic beats in 24 hours, or >2% of total beats.
    * Ventricular tachycardia (ventricular tachycardia defined as ≥ 3 successive ventricular ectopic beats at a rate of > 120 bpm).
    * Abnormal T-wave morphology.
    * QT interval corrected using the Fridericia's formula (QTcF) > 450 ms at screening. Participant with borderline deviations (within 10% of upper limit) from these criteria may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.
15. Has vital signs outside of the following normal range at screening, Day -1, or

    Day 1 pre-dose:

    - Blood pressure (BP):

    Supine BP (after at least 5 minutes of supine rest):
    * Systolic blood pressure: 90 - 140 mmHg.
    * Diastolic blood pressure: 40 - 90 mmHg. - Supine pulse rate after at least 5 minutes of rest: 45 - 90 bpm. At the discretion of the PI, the 24-hour Holter, in addition to the screening vital signs, may be used to assess the resting heart rate.
16. Signs and/or symptoms of a clinically relevant acute illness in the four-week period prior to screening.
17. Veins unsuitable for intravenous puncture or cannulation on either arm (e.g., veins that are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture).
18. Known hypersensitivity to any medicines administered in the trial, including quinolone-class antibiotics.
19. Unless approved explicitly by the PI, use of any prescription medications within 7 days or 10 half-lives (whichever is longer) prior to Day 1, or any over the counter (OTC) medication (including multivitamin, herbal, or homeopathic preparations, excluding hormonal contraception, hormone replacement therapy, and/or paracetamol- maximum 2g per day) within 7 days prior to Day 1 of the dosing period. Medicines predisposing to lactic acidosis, such as inhaled salbutamol, should not be used for the duration of the dosing period.
20. Administration of antibiotics 7 days prior to the admission for the study or plan to take antibiotics during the study.
21. Treatment with an investigational drug within 90 days prior to admission or having participated in more than three investigational drug studies within one year prior to admission.
22. Unless approved explicitly by the PI, positive test results for alcohol or drugs of abuse at screening and on Day -1.
23. Female participants who are pregnant (including a positive serum pregnancy test at screening and on Day-1) or breastfeeding.
24. Presence or history of drug or alcohol abuse in the last 5 years, or inability to refrain from alcohol use from 48 hours before screening, dosing, and each scheduled visit until the end of the study. Alcohol abuse is defined as regular weekly intake of more than 14 units (for both males and females), using the following NHS alcohol tracker http://www.nhs.uk/Tools/Pages/drinkstracker. aspx.
25. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine containing products in any form (e.g., gum, patch, electronic cigarettes) within 1 month prior to the planned first day of dosing.
26. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
27. Has a legal or mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the study requirements at screening.
28. Any circumstances or conditions, which, in the opinion of the Investigator, may affect full participation in the study or compliance with the protocol.
29. An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
30. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), participation, or enrolment in this study. Participants who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved.
31. Abstain from blood and plasma donation during the study and up to 3 months after completion of the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinically significant ECG morphology and interval changes from baseline | Specified timepoints for 4 days and at follow up visit on Day10-D17
  ECG Analysis Mean QT/QTc values will be calculated for each time point (triplicate ECG) for subsequent analyses. Telemetry data gathered during the study may be used in the optional exploratory analysis of drug related QT/QTc interval changes.
  The primary baseline corrections will be calculated using averaged QTc pre-dose baseline values (three pre-dose time points). This single value will be used to calculate ΔQTc. A supplementary analysis to calculate ΔΔQTc may be performed using pooled placebo data. The effect on QTc will be calculated using concentration-effect analysis based on the placebo-corrected change from average baseline.
Cardiac intervals/subintervals calculated using concentration-effect analysis on Days 1, 2, and 3. | Specified timepoints for 3 days
  The primary baseline corrections will be calculated using averaged QTc pre-dose baseline values (three pre-dose time points). This single value will be used to calculate ΔQTc. A supplementary analysis to calculate ΔΔQTc may be performed using pooled placebo data. The effect on QTc will be calculated using concentration-effect analysis based on the placebo-corrected change from average baseline.
The paired PK of blood glucose and moxifloxacin (Cmax) | 4 Days
  PK parameter: Maximum observed plasma concentration (Cmax)
  * Glucose
    * Day 1: Cmax
    * Day 2: Cmax
    * Day 3: Cmax
    * Day 4: Cmax
  * Moxifloxacin
    * Day 3: Cmax
    * Day 4: Cmax
The paired PK of blood glucose and moxifloxacin (Tmax) | 4 days
  PK parameter:
  time to reach maximum plasma concentration (Tmax)
  * Glucose
    * Day 1: Tmax
    * Day 2: Tmax
    * Day 3: Tmax
    * Day 4: Tmax
  * Moxifloxacin
    * Day 3: Tmax
    * Day 4: Tmax
The paired PK of blood glucose and moxifloxacin (AUC) | 4 days
  PK parameter: Area under the plasma concentration-time curve (AUC).
  * Glucose
    * Day 1: AUC
    * Day 2: AUC
    * Day 3: AUC
    * Day 4: AUC
  * Moxifloxacin
    * Day 3: AUC
    * Day 4: AUC
Cardiac interval/subinterval parameters | 4 days
  Cardiac interval/subinterval parameters (QTcF, JTpc, TpTe) prior to glucose administration compared to post-administration

SECONDARY OUTCOMES:
Comparison of the PK of blood glucose and moxifloxacin with cardiac interval/subinterval parameters and ECG morphology between sexes on Days 1, 2, 3 and 4 | Specified time points over 4 days
  Comparison between males and females of the paired PK blood glucose and moxifloxacin, and cardiac interval/subinterval parameters (QTcF, JTpc, TpTe) prior to glucose administration compared to post-administration. PK parameters include maximum observed plasma concentration (Cmax), time to reach maximum plasma concentration (tmax), area under the plasma concentration-time curve (AUC).
  * Glucose
    * Day 1: Cmax, tmax, AUC
    * Day 2: Cmax, tmax, AUC
    * Day 3: Cmax, tmax, AUC
    * Day 4: Cmax, tmax, AUC
  * Moxifloxacin
    * Day 3: Cmax, tmax, AUC
    * Day 4: Cmax, tmax, AUC
  * QTcF, JTpc, TpTe o Days 1, 2, and 3.
• Concentration effect analysis between male and female volunteers on Days 1, 2, 3 and 4 | specified timepoints over 4 days
  Comparison of males vs females of the primary baseline corrections calculated using averaged QTc pre-dose baseline values (three pre-dose time points). This single value will be used to calculate ΔQTc. A supplementary analysis to calculate ΔΔQTc may be performed using pooled placebo data. The effect on QTc will be calculated using concentration-effect analysis based on the placebo-corrected change from average baseline.
The incidence of treatment-emergent adverse events (TEAEs) | From screening to follow up approximately 75 days
  Proportion of participants with clinically significant changes in laboratory safety tests (haematology, chemistry, coagulation and urinalysis), proportion of participants with morphological and/or rhythm abnormalities on ECG, proportion of participants with clinically significant changes in ECG time intervals (PR, QRS, QT and QTc intervals) and proportion of participants with clinically significant changes in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate and tympanic temperature).

OTHER OUTCOMES:
To gain a comprehensive understanding of the molecular factors driving differences between male and female participants, by analysing a set of relevant biomarkers: insulin, C-peptide and glucagon. | 3 days
  Change from baseline for individual biomarkers over time, correlated with changes in blood glucose and QTc interval parameters, ECG morphology and concentration effect analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided